CLINICAL TRIAL: NCT02373163
Title: Characterization of Arterial Hypertension and Efficacy of Blood-pressure Lowering Therapy at Different Altitudes Above Sea Level
Brief Title: INTERVENCION Trial
Acronym: INTERVENCION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prevencion (Other)
Responsible Party: Principal Investigator, Josefina Medina-Lezama, MD, Principal Investigator, Prevencion
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INTERVENCION Trial
Record Dates: First submitted 2015-02-10; First posted 2015-02-26 (Estimated); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Blood Pressure, High
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide; Amlodipine; Telmisartan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diuretic (Active Comparator): Therapy with hydrochlorothiazide (25 mg daily) taken once daily between 6 and 8 AM
  Interventions: Drug: Hydrochlorothiazide
- Calcium-channel blocker (Active Comparator): Therapy with amlodipine (10 mg daily) taken once daily between 6 and 8 AM
  Interventions: Drug: Amlodipine
- Angiotensin Receptor Blocker (Active Comparator): Therapy with Telmisartan (80 mg daily) taken once daily between 6 and 8 AM
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Hydrochlorothiazide — Arm: Active Comparator: Diuretic Therapy with hydrochlorothiazide (25 mg daily) taken once daily between 6 and 8 AM Arm: Active Comparator: Calcium-channel blocker Therapy with amlodipine (10 mg daily) taken once daily between 6 and 8 AM Arm: Active Comparator: Angiotensin Receptor Blocker Therapy with Telmisartan (80 mg daily) taken once daily between 6 and 8 AM
  Other Names: HCTZ
  Arms: Diuretic
Drug: Amlodipine — Therapy with amlodipine (10 mg daily) taken once daily between 6 and 8 AM
  Arms: Calcium-channel blocker
Drug: Telmisartan — Therapy with Telmisartan (80 mg daily) taken once daily between 6 and 8 AM
  Arms: Angiotensin Receptor Blocker

SUMMARY:
This trial is designed to:

1. Assess the response to montherapy with : a thiazide diuretic (HCTZ), a calcium-channel blocker (CCB, amlodipine) and an angiotensin-receptor blocker (telmisartan), among hypertensive subjects who live at sea level, at medium altitude above sea level and at high altitude above sea level.
2. To test whether diferentes exist in the response to therapy among subjects who live at different altitude above sea level
3. To assess the hemodynamic characteristics of hypertension in populations that live at sea level, at medium altitude above sea level, and at high altitude above sea level.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45-75 years. Enrollment will be stratified by age group (50-65 and 66-80 years), gender and altitude above sea level
2. Leaving in the enrollment cities for at least 2 years
3. Untreated hypertension for at least 2 weeks
4. Systolic BP between 140 and 160 mmHg and/or diastolic BP between 90 and 99 mmHg, in the absence of therapy.

Exclusion Criteria:

1. Diabetes mellitus.
2. Chronic kidney disease (estimated glomerular filtration rate <60 ml / minute / 1.73 m2 of body surface area.
3. Smoking.
4. Lung disease, liver disease or active cancer
5. Any factor that, in the opinion of the investigator, decreases short-term survival
6. Psychiatric illness
7. Inability to provide informed consent
8. Established heart disease (previous myocardial infarction, heart failure, valvular heart disease, cardiomyopathy, atrial fibrillation or any significant cardiac arrhythmia)
9. History of cerebrovascular disease
10. History of orthostatic hypotension.
11. History of syncope.
12. History of allergy of adverse effects to study medications or drugs of the same pharmacologic classes.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Investigacion PREVENCION, Arequipa, AQP, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Medina-Lezama J, Zea-Diaz H, Morey-Vargas OL, Bolanos-Salazar JF, Postigo-Macdowall M, Paredes-Diaz S, Corrales-Medina F, Valdivia-Ascuna Z, Cuba-Bustinza C, Villalobos-Tapia P, Munoz-Atahualpa E, Chirinos-Pacheco J, Raij L, Chirinos JA. Prevalence and patterns of hypertension in Peruvian Andean Hispanics: the PREVENCION study. J Am Soc Hypertens. 2007 May-Jun;1(3):216-25. doi: 10.1016/j.jash.2007.02.003. PMID 20409853

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diuretic | Calcium-channel Blocker | Angiotensin Receptor Blocker
Started | 56 | 55 | 55
Completed | 56 | 55 | 55
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diuretic | Calcium-channel Blocker | Angiotensin Receptor Blocker | Total
Number analyzed (Participants) | 56 | 55 | 55 | 166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 35 | 36 | 104
  >=65 years | 23 | 20 | 19 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.32 (10.06) | 60.95 (8.35) | 60.38 (8.41) | 59.87 (9.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 29 | 86
  Male | 28 | 26 | 26 | 80
Region of Enrollment [Number; unit: participants]
  Peru | 56 | 55 | 55 | 166
Systolic blood pressure, office [Mean (Standard Deviation); unit: mm Hg] | 144.68 (9.63) | 143.62 (9.52) | 146.2 (10.59) | 144.83 (9.92)
Diastolic blood pressure, office [Mean (Standard Deviation); unit: mm Hg] | 84.41 (7.27) | 86.7 (12.01) | 86.38 (8.63) | 85.82 (9.50)
24-hour Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 127.98 (10.80) | 126.80 (10.65) | 128.40 (14.69) | 127.73 (12.13)
24-hour Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 78.22 (7.90) | 77.43 (9.56) | 78.52 (9.78) | 78.06 (9.07)
24-hour Mean Arterial Pressure [Mean (Standard Deviation); unit: mm Hg] | 101.02 (8.28) | 100.04 (9.29) | 101.37 (10.93) | 100.81 (9.51)
24-hour Pulse Pressure [Mean (Standard Deviation); unit: mm Hg] | 49.76 (8.60) | 49.37 (7.87) | 49.88 (11.15) | 49.67 (9.26)
Carotid Pulse Pressure [Mean (Inter-Quartile Range); unit: mm Hg] | 53.50 [44.75 to 61.00] | 53.00 [41.50 to 63.00] | 55.00 [45.00 to 61.00] | 54.00 [43.25 to 61.75]
Carotid-Femoral Pulse Wave Velocity [Mean (Inter-Quartile Range); unit: meters/second] | 8.70 [7.15 to 10.10] | 8.20 [7.30 to 9.95] | 8.35 [6.82 to 10.45] | 8.40 [7.10 to 10.10]

OUTCOME MEASURES:

1. Primary Outcome: Change is 24-hour Systolic Blood Pressure From Baseline to 4 Weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Diuretic | Calcium-channel Blocker | Angiotensin Receptor Blocker
Number analyzed (Participants) | 56 | 55 | 55
mmHg | -5.9 (8.4) | -7.5 (9.2) | -8.4 (8.8)

2. Secondary Outcome: Change in 24-hour Diastolic Blood Pressure From Baseline to 4 Weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Diuretic | Calcium-channel Blocker | Angiotensin Receptor Blocker
Number analyzed (Participants) | 56 | 55 | 55
mmHg | -3.5 (5.7) | -4.7 (5.5) | -5.6 (6.2)

3. Secondary Outcome: Change in 24-hour Mean Arterial Pressure From Baseline to 4 Weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Diuretic | Calcium-channel Blocker | Angiotensin Receptor Blocker
Number analyzed (Participants) | 56 | 55 | 55
mmHg | -4.6 (6.5) | -6.0 (6.9) | -6.9 (7.1)

4. Secondary Outcome: Change in 24 Hour Pulse Pressure From Baseline to 4 Weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Diuretic | Calcium-channel Blocker | Angiotensin Receptor Blocker
Number analyzed (Participants) | 56 | 55 | 55
mmHg | -2.4 (5.4) | -2.8 (5.6) | -2.8 (4.9)

5. Secondary Outcome: Change in Central (Aortic) Pulse Pressure, Carotid Arterial, From Baseline to 4 Weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Diuretic | Calcium-channel Blocker | Angiotensin Receptor Blocker
Number analyzed (Participants) | 56 | 55 | 55
mmHg | -11.6 (15.6) | -9.6 (18.7) | -11.2 (14.2)

6. Secondary Outcome: Change in Carotid-femoral Pulse Wave Velocity From Baseline to 4 Weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Diuretic | Calcium-channel Blocker | Angiotensin Receptor Blocker
Number analyzed (Participants) | 56 | 55 | 55
m/sec | -0.4 (1.3) | -0.3 (1.3) | -0.6 (2.0)

ADVERSE EVENTS:
Arm/Group | Diuretic | Calcium-channel Blocker | Angiotensin Receptor Blocker
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/56 | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No